CLINICAL TRIAL: NCT06972628
Title: 177Lu-PSMA-617 (Pluvicto) for the Treatment of Patients With Progressive PSMA-Positive Metastatic Castration-Resistant Prostate Cancer (mCRPC) and Super Scan Bone Scan
Brief Title: Treatment of Patients With Progressive mCRPC With 177Lu-PSMA-617
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ebrahim S Delpassand (Other)
Responsible Party: Sponsor-Investigator, Ebrahim S Delpassand, Chairman & Medical Director, Excel Diagnostics & Nuclear Oncology Center, Excel Diagnostics and Nuclear Oncology Center
Organization: Excel Diagnostics and Nuclear Oncology Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Super-Lu-177
Record Dates: First submitted 2025-04-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer; Prostate Cancer Patients With Bone Metastasis; Prostate Cancer (CRPC); Prostate Cancer; Prostate Cancer Metastatic
Keywords: Metastatic Castration-Resistant Prostate Cancer (mCRPC); super scan bone scan; Prostate Cancer patients with bone metastasis; prostate cancer (CRPC); Prostate cancer; Prostate cancer metastatic
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Intervention Model Description: This study uses an FDA-approved drug (PLUVICTO). Therefore, it is not subject to phase categorization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Administering Lutetium-177-PSMA-617 (PLUVICTO)

INTERVENTIONS:
Drug: Administering Lutetium-177-PSMA-617 (PLUVICTO) — The study begins with a first cohort of three participants, each receiving a dose of 100 millicuries (mCi). After administration, participants are monitored for any dose-limiting toxicities (DLTs) during a predefined observation window. If fewer than two participants experience a DLT in a given cohort, the dose will be escalated for the next group. The dose escalation schedule is structured as follows: the second cohort receives 130 mCi (a 30% increase), the third cohort receives 162.5 mCi (a 25% increase), and the fourth cohort receives 200 mCi, a dose that is already FDA-approved and clinically accepted for mCRPC. This stepwise escalation continues until the 200 mCi dose is reached, or until two or more DLTs are observed in any cohort. If that occurs, escalation stops immediately, and the maximum tolerated dose is considered to be the previous lower dose. This becomes the optimal tolerated dose (OTD). After identifying the OTD, additional participants will be enrolled for treatment.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Lutetium-177-PSMA-617 (PLUVICTO) in patients with metastatic castration-resistant prostate cancer (mCRPC) and extensive bone metastases, which appear as a "super scan" pattern on a bone scan.

Pluvicto is FDA-approved, but patients with super scan bone scans were previously excluded from the VISION clinical trial, leaving a knowledge gap.

The study will enroll up to 30 men with metastatic castration-resistant prostate cancer, with an initial dosing approach that differs from the standard dose.

The safety and tolerability of PLUVICTO will be evaluated in this study, with a focus on identifying the optimal dose for this population.

This study addresses an important gap in understanding how Pluvicto performs in mCRPC patients with super scan findings.

DETAILED DESCRIPTION:
This clinical study investigates the safety and effectiveness of the FDA-approved drug Pluvicto (Lu-177-PSMA617).

It focuses on a unique group of patients with metastatic castration-resistant prostate cancer (mCRPC) who present with a "super scan" on bone scintigraphy-a pattern indicating widespread cancer in the bones.

These patients were excluded from prior trials like the VISION study, leaving a critical gap in clinical understanding.

The trial aims to identify the optimal safe dose of Pluvicto using a modified 3+3 dose-escalation method, beginning at a low dose that increases, and eventually reaching up to 200 mCi.

Participants will receive a total of six doses, spaced every 6 ± 1 weeks. Primary objectives include determining the maximum tolerated dose and monitoring safety using CTCAE version 5.0 criteria.

Efficacy will be evaluated through PSA level reductions based on PCWG3 guidelines.

Secondary endpoints include quality of life, radiologic response (RECIST v1.1), and overall survival.

Exploratory endpoints involve PSMA PET/CT imaging to measure treatment response through SUVmean and lesion changes.

The study includes up to 30 participants and will include expanded enrollment once the optimal dose is determined.

Routine lab tests (CBC, CMP, PSA, testosterone) and patient-reported side effects will be monitored throughout the study.

Long-term follow-up for survival and safety will continue every six months for up to five years.

Imaging (CT/MRI, bone scans, and optional PET/CT) will be performed at baseline, mid-treatment, end of treatment, and every three months post-treatment.

A complete or partial response, stable disease, or progression will be defined using both RECIST and PCWG3 guidelines.

Monthly PSA checks will continue for up to 24 months or until disease progression.

PLUVICTO is administered via IV infusion over 2-5 minutes during each session. Participants may discontinue due to progression, intolerable side effects, non-compliance, or other clinical decisions.

This study is essential in determining how to safely extend Pluvicto therapy to a previously unstudied and high-risk patient group.

Its results may expand access to this radioligand therapy and guide future treatment decisions in prostate cancer care.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign an informed consent form (ICF).
2. Willingness and ability to comply with study requirements.
3. Age ≥18 years.
4. Presence of skeletal metastases with a superscan pattern on a 99mTc-MDP/HDP bone scan, defined by significantly increased skeletal radioisotope uptake relative to soft tissues and faint or absent renal activity.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. Hemoglobin ≥9.0 g/dL.
7. Platelet count ≥90 × 10⁹/L.
8. White blood cell count ≥2.0 × 10⁹/L, absolute neutrophil count (ANC) >1.5 × 10⁹/L.

   o These hematologic criteria must be met without recent transfusions (within 28 days prior to the first study treatment) or growth factor support (within 21 days).
9. Serum/plasma creatinine ≤1.5 × upper limit of normal (ULN).
10. Histological, pathological, or cytological confirmation of prostate cancer.
11. Positive PSMA PET/CT scan showing at least one PSMA-positive metastatic lesion.
12. Castrate-level serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L).
13. Prior treatment with at least one androgen receptor-axis-targeted therapy (ARAT).

Exclusion Criteria:

1. Prior treatment with radiopharmaceuticals (e.g., Strontium-89, Samarium-153, Rhenium- 186, Rhenium-188, Radium-223, hemi-body irradiation) within six months before start of treatment under this protocol.
2. Prior PSMA-targeted radioligand therapy.
3. Systemic anti-cancer therapy (e.g., chemotherapy, immunotherapy, monoclonal antibodies) within four weeks before screening visit.
4. Known hypersensitivity to PLUVICTO or its components.
5. Concurrent treatment with other cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
6. Renal impairment (estimated glomerular filtration rate <60 mL/min), hemoglobin <9 g/dL, ANC <1.5 × 10⁹/L, or platelets < 90 × 10⁹/L.
7. History of CNS metastases unless treated and stable for 6 months, with no ongoing corticosteroid use.
8. Symptomatic or impending spinal cord compression.
9. Other malignancies impacting life expectancy or interfering with study assessments. Exceptions include non-melanoma skin cancer or superficial bladder cancer that has been adequately treated.
10. Major surgery within 30 days prior to enrollment.
11. Plans to conceive or father a child during treatment and up to six months post-treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-23 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival | From date of enrollment until the date of first documented radiographic disease progression or date of death from any cause, whichever came first, assessed up to 24 months.
  rPFS: Defined as the time from enrollment to radiographic disease progression, based on Prostate Cancer Working Group 3 (PCWG3) Guidelines (Scher et al., 2016), or death from any cause.
Overall Survival | From date of enrollment until the date of death from any cause, assessed up to 24 months.
  OS: Defined as the time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim S. Delpassand, M.D. Chairman & Medical Director, MD., Nuclear Medicine, Principal Investigator — Excel Diagnostics & Nuclear Oncology Center
Locations (1):
- Excel Diagnostics & Nuclear Oncology Center, Houston, Texas, United States

REFERENCES:
- [Background] Hartrampf PE, Weinzierl FX, Buck AK, Rowe SP, Higuchi T, Seitz AK, Kubler H, Schirbel A, Essler M, Bundschuh RA, Werner RA. Matched-pair analysis of [177Lu]Lu-PSMA I&T and [177Lu]Lu-PSMA-617 in patients with metastatic castration-resistant prostate cancer. Eur J Nucl Med Mol Imaging. 2022 Jul;49(9):3269-3276. doi: 10.1007/s00259-022-05744-6. Epub 2022 Mar 4. PMID 35243517
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Banerjee SR, Pullambhatla M, Byun Y, Nimmagadda S, Green G, Fox JJ, Horti A, Mease RC, Pomper MG. 68Ga-labeled inhibitors of prostate-specific membrane antigen (PSMA) for imaging prostate cancer. J Med Chem. 2010 Jul 22;53(14):5333-41. doi: 10.1021/jm100623e. PMID 20568777
- [Background] Hope TA, Abbott A, Colucci K, Bushnell DL, Gardner L, Graham WS, Lindsay S, Metz DC, Pryma DA, Stabin MG, Strosberg JR. NANETS/SNMMI Procedure Standard for Somatostatin Receptor-Based Peptide Receptor Radionuclide Therapy with 177Lu-DOTATATE. J Nucl Med. 2019 Jul;60(7):937-943. doi: 10.2967/jnumed.118.230607. PMID 31263080
- [Background] Ahmadzadehfar H, Eppard E, Kurpig S, Fimmers R, Yordanova A, Schlenkhoff CD, Gartner F, Rogenhofer S, Essler M. Therapeutic response and side effects of repeated radioligand therapy with 177Lu-PSMA-DKFZ-617 of castrate-resistant metastatic prostate cancer. Oncotarget. 2016 Mar 15;7(11):12477-88. doi: 10.18632/oncotarget.7245. PMID 26871285
- [Background] Messiou C, Cook G, deSouza NM. Imaging metastatic bone disease from carcinoma of the prostate. Br J Cancer. 2009 Oct 20;101(8):1225-32. doi: 10.1038/sj.bjc.6605334. Epub 2009 Sep 29. PMID 19789531
- [Background] Caglar M, Tuncel M, Yildiz E, Karabulut E. Bone scintigraphy as a gatekeeper for the detection of bone metastases in patients with prostate cancer: comparison with Ga-68 PSMA PET/CT. Ann Nucl Med. 2020 Dec;34(12):932-941. doi: 10.1007/s12149-020-01529-9. Epub 2020 Sep 25. PMID 32975741
- [Background] Askari E, Shakeri S, Roustaei H, Fotouhi M, Sadeghi R, Harsini S, Vali R. Superscan Pattern on Bone Scintigraphy: A Comprehensive Review. Diagnostics (Basel). 2024 Oct 6;14(19):2229. doi: 10.3390/diagnostics14192229. PMID 39410633
- [Background] Manov JJ, Roth PJ, Kuker R. Clinical Pearls: Etiologies of Superscan Appearance on Fluorine-18-Fludeoxyglucose Positron Emission Tomography-Computed Tomography. Indian J Nucl Med. 2017 Oct-Dec;32(4):259-265. doi: 10.4103/ijnm.IJNM_56_17. PMID 29142340
- [Background] Manohar PR, Rather TA, Khan SH, Malik D. Skeletal Metastases Presenting as Superscan on Technetium 99m Methylene Diphosphonate Whole Body Bone Scintigraphy in Different Type of Cancers: A 5-Year Retro-prospective Study. World J Nucl Med. 2017 Jan-Mar;16(1):39-44. doi: 10.4103/1450-1147.181153. PMID 28217018
- See also: Data on file. VISION [PSMA-617-01] study. Novartis Pharmaceuticals Corp; 2021. — https://us.pluvicto.com/about-mcrpc?site=FA-11346005-FA-11346011GK101501&utm_source=google&utm_mlr=FA-11346005-FA-11346011&utm_medium=cpc&utm_campaign=google_branded_pluvicto-dtc-branded-phrase-fa-11346005-fa-11346011%3Bs%3Bph%3Bbr%3Bonc%3Bdtc%3Bbr_apr-2025&utm_content=plu_prostate-cancer_kw_n2_indication-psma&utm_term=psma%20lutetium%20177&gad_source=1&gbraid=0AAAAAoJ1MW4V9ow_tIT2i_8_D6jCD5_n-&gclid=EAIaIQobChMIt_Po-NzGjAMVL1N_AB1ALBMQEAAYASAAEgLrsPD_BwE&gclsrc=aw.ds
- See also: American Cancer Society . Cancer Facts and Statistics: American Cancer Society. 2015 — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2015.html